CLINICAL TRIAL: NCT06394934
Title: Impact of Home and Clinical Blood Pressure Variability on Arteriosclerosis and Metabolic Indicators
Brief Title: Home Blood Pressure Variability and Its Link to Arteriosclerosis and Metabolic Dysfunction in Hypertensive Patients
Status: Recruiting | Type: Observational
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Korean Society of Hypertension (Other)
Responsible Party: Principal Investigator, Hyung Joon Joo, Professor, Korea University Anam Hospital
Other Study IDs: HBPV-ARTMET-2023
Record Dates: First submitted 2024-04-21; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Hypertension; Blood Pressure Monitoring, Home; Arteriosclerosis; Metabolic Syndrome X
Keywords: Home Blood Pressure Monitoring; Blood Pressure Variability; Pulse Wave Velocity; Arteriosclerosis
MeSH Terms: conditions — Hypertension; Arteriosclerosis; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Home BP Monitoring Cohort: Participants in this cohort are hypertensive adults who will use the Healthscan mobile application to monitor and record their blood pressure at home.
  Interventions: Behavioral: Healthscan App

INTERVENTIONS:
Behavioral: Healthscan App — Participants will use the Healthscan mobile application to monitor and record their daily blood pressure at home. The app allows participants to enter their BP measurements, which are then used to calculate blood pressure variability (BPV). The app's use is intended as a non-invasive, practical tool for patient self-management and longitudinal health monitoring in hypertensive individuals.

SUMMARY:
This observational study investigates the correlation between home blood pressure variability (BPV) and arteriosclerosis, alongside metabolic indicators, in hypertensive patients over a three-year period. The research specifically focuses on the predictive value of home BPV for major adverse cardiovascular events (MACE) including myocardial infarction, stroke, and heart failure hospitalizations. Utilizing a mobile application called Healthscan for daily BP monitoring, the study aims to enhance the understanding of how BPV impacts cardiovascular and metabolic health in a real-world setting.

DETAILED DESCRIPTION:
Objective:

This longitudinal, non-randomized study aims to explore the prognostic value of home-measured blood pressure variability (BPV) in predicting arteriosclerosis and metabolic dysfunction in patients with hypertension. By examining the relationship between home BPV and several vascular and metabolic health indicators, this study seeks to validate home BP monitoring as a crucial component of hypertension management.

Study Design:

Participants will be recruited from multiple clinical settings and followed for a three-year period, during which they will use the Healthscan mobile application to record their daily blood pressure readings. The primary outcome measure is the correlation between home BPV and pulse wave velocity, a key marker of arteriosclerosis. Secondary outcomes include other arteriosclerosis indicators such as ankle-brachial index and central systolic blood pressure, as well as metabolic indicators like fasting glucose and lipid profiles.

Methodology:

Approximately 4,188 hypertensive patients over 19 years old, with a history of antihypertensive medication use, will be enrolled. Data collection will be facilitated through the Healthscan app, which participants will use to enter their BP measurements. This data will provide insights into the average blood pressure and variability over specified periods. The study will utilize Pearson or Spearman correlation coefficients to assess the relationships between home BPV and health indicators, with multivariate regression models adjusting for potential confounders.

Ethical Considerations:

The study has been approved by an institutional review board and all participants will provide written informed consent. The study prioritizes data confidentiality and participant privacy, with data being securely stored and managed.

Significance:

By correlating BPV with arteriosclerosis and metabolic parameters, the study could significantly impact clinical practices by reinforcing the role of home BP monitoring in the early detection and management of cardiovascular risks in hypertensive patients. This could potentially lead to more personalized and effective healthcare strategies, ultimately improving patient outcomes in hypertension management.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years or older.
2. Diagnosed with hypertension.
3. Regular use of antihypertensive medication for at least two years.
4. Access to a home blood pressure monitor.
5. Comprehensive medical records available for the past year.

Exclusion Criteria:

1. Participants who are unable to consent or who might not reliably use the home monitoring app.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult hypertensive patients from various clinical settings, including community clinics and academic hospitals. Participants are broadly recruited to reflect a diverse population regarding age, sex, and severity of hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 4188 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between Home Blood Pressure Variability and Pulse Wave Velocity | 1 year
  Measure the strength and nature of the relationship between variability in home-monitored blood pressure and pulse wave velocity, a primary indicator of arteriosclerosis.

SECONDARY OUTCOMES:
Association between Home BPV and Additional Arteriosclerosis Indicators | 1 year
  Assess the correlation of home BPV with other arteriosclerosis indicators including ankle-brachial index, central systolic blood pressure, and second systolic peak blood pressure.
Correlation between Home BPV and Metabolic Indicators | 1 year
  Evaluate the association between home BPV and metabolic health indicators such as fasting glucose levels and lipid profiles (total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides).

OTHER OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) | 3 years
  Monitor and record the incidence of major adverse cardiovascular events including myocardial infarction, stroke, and heart failure hospitalizations among study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Joon Joo, MD PhD, Principal Investigator — Korea University Anam Hospital
Locations (2):
- South Korea (2):
  - Korea University Anam Hospital, Seoul
  - Korea Univeristy Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided
As of now, the decision to share individual participant data (IPD) from this study remains undecided. We recognize the potential value of sharing data to advance scientific knowledge and improve patient care; however, we also prioritize the privacy and confidentiality of our participants. Our final decision will be informed by a comprehensive risk-benefit analysis, ensuring any data-sharing complies with all applicable privacy laws and ethical guidelines. We commit to updating this plan once a conclusive decision has been made, based on these detailed evaluations and consultations.

REFERENCES:
- [Background] Parati G, Torlasco C, Pengo M, Bilo G, Ochoa JE. Blood pressure variability: its relevance for cardiovascular homeostasis and cardiovascular diseases. Hypertens Res. 2020 Jul;43(7):609-620. doi: 10.1038/s41440-020-0421-5. Epub 2020 Mar 13. PMID 32203448
- [Background] Rosei EA, Chiarini G, Rizzoni D. How important is blood pressure variability? Eur Heart J Suppl. 2020 Jun;22(Suppl E):E1-E6. doi: 10.1093/eurheartj/suaa061. Epub 2020 Apr 6. PMID 32523429
- [Background] Johansson JK, Niiranen TJ, Puukka PJ, Jula AM. Prognostic value of the variability in home-measured blood pressure and heart rate: the Finn-Home Study. Hypertension. 2012 Feb;59(2):212-8. doi: 10.1161/HYPERTENSIONAHA.111.178657. Epub 2012 Jan 3. PMID 22215704
- [Background] Juhanoja EP, Niiranen TJ, Johansson JK, Puukka PJ, Jula AM. Agreement between ambulatory, home, and office blood pressure variability. J Hypertens. 2016 Jan;34(1):61-7. doi: 10.1097/HJH.0000000000000772. PMID 26630214
- [Background] Ntineri A, Kalogeropoulos PG, Kyriakoulis KG, Aissopou EK, Thomopoulou G, Kollias A, Stergiou GS. Prognostic value of average home blood pressure and variability: 19-year follow-up of the Didima study. J Hypertens. 2018 Jan;36(1):69-76. doi: 10.1097/HJH.0000000000001497. PMID 28777132
- [Background] Whelton PK, Carey RM, Mancia G, Kreutz R, Bundy JD, Williams B. Harmonization of the American College of Cardiology/American Heart Association and European Society of Cardiology/European Society of Hypertension Blood Pressure/Hypertension Guidelines: Comparisons, Reflections, and Recommendations. Circulation. 2022 Sep 13;146(11):868-877. doi: 10.1161/CIRCULATIONAHA.121.054602. Epub 2022 Aug 11. PMID 35950927
- [Derived] Yu HY, Cha JJ, Cho DH, Kim MN, Oh SW, Park JH, Cho KH, Shin SY, Kim EJ, Joo HJ. Impact of home and clinical blood pressure variability on arteriosclerosis and metabolic indicators: a prospective multicenter registry study. Clin Hypertens. 2025 Nov 1;31:e37. doi: 10.5646/ch.2025.31.e37. eCollection 2025. PMID 41209073